CLINICAL TRIAL: NCT01468649
Title: Phase II Real-Time NIR-Guided Sentinel Lymph Node Mapping in Breast Cancer
Brief Title: Real-Time Near-infrared (NIR) Mapping of Sentinel Lymph Nodes in Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Brigham and Women's Hospital (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, John V. Frangioni, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2007P000431
Record Dates: First submitted 2011-06-30; First posted 2011-11-09 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Sentinel Lymph Node Mapping; Intraoperative Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast Cancer SLN Mapping (Experimental): Fifty participants consented who will be undergoing standard of care for breast cancer SLN mapping with Tc-99m will be enrolled in this study.
  Interventions: Device: NIR Imaging with FLARE and Mini-FLARE Imaging System

INTERVENTIONS:
Device: NIR Imaging with FLARE and Mini-FLARE Imaging System — A custom-designed imaging platform that utilizes NIR fluorescence optics will be employed to identify the injected dye and its path through the lymphatic track, and its eventual highlighting of the SLN. Both color images and NIR images will be merged to give the operating surgeon a clear picture of the ICG track superimposed over anatomical landmarks. This technique will identify the SLN and provide an accurate video image of its location.
  Other Names: Fluorescence assisted imaging

SUMMARY:
The objective of this Phase II study is to assess the diagnostic accuracy of sentinel lymph node (SLN) identification in patients with breast cancer using near-infrared (NIR) fluorescence optical imaging.

DETAILED DESCRIPTION:
Fifty participants consented from Brigham and Women's Hospital (currently enrolling) and Beth Israel Deaconess Medical Center (currently non-enrolling), who will be undergoing standard of care for breast cancer SLN mapping with Tc-99m will be enrolled in this study.

Prior to surgery, patients will undergo lymphoscintigraphy as is standard of care. At the time of SLN mapping, the patient will be injected with indocyanine green dye (ICG). Concurrently, a custom-designed imaging platform that utilizes NIR fluorescence optics will be employed to identify the dye and its path through the lymphatic track, and its eventual highlighting of the SLN. Both color images and NIR images will be merged to give the operating surgeon a clear picture of the ICG track superimposed over anatomical landmarks. This technique will identify the SLN and provide an accurate video image of its location. The surgeon will resect all SLNs identified by Tc-99m or NIR fluorescence, and then confirm the radioactivity and NIR fluorescence signal in each after resection.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have histologically confirmed breast cancer and be deemed an appropriate surgical candidate with consent for a sentinel lymph node mapping by their oncologic surgeon.
* Age minimum: 18 years.
* Participant must be receiving a planned lymphoscintigraphy procedure.
* Participant must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who choose not to proceed with sentinel lymph node biopsy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to indocyanine green, including those patients with a history of iodide or seafood allergy.
* Women who are pregnant or may become pregnant, as well as those women who are breastfeeding, will be excluded from this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity of Real-Time Intraoperative NIR Mapping | One Day (day 1)
  To determine the sensitivity of real-time intraoperative NIR lymphatic mapping in the identification of the sentinel lymph node in human breast cancer as compared to the standard of care, Technicium 99 (Tc-99).

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | One Day (day 1)
  To evaluate the incidence of significant adverse reactions due to both NIR lymphatic mapping and indocyanine green.

CONTACTS AND LOCATIONS:
Overall Officials: John V. Frangioni, M.D., Ph.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States